CLINICAL TRIAL: NCT04974476
Title: A Comparison of Onsite vs. Virtual Fitness Program on Anthropometric Measures, Aerobic Fitness, and Vascular Markers of Cardiac Risk Markers in Overweight/Obese Premenopausal Women
Brief Title: Onsite vs. Virtual Group Fitness in Overweight/Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Arlette Perry, Professor, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20210038
Record Dates: First submitted 2021-07-14; First posted 2021-07-23 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Overweight and Obesity
Keywords: Exercise Program
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-person exercise training group (Experimental): participants in this group will receive in person exercise HIIT training 3 days a week for 12 weeks
  Interventions: Other: HIIT Exercise Training
- Virtual exercise training group (Experimental): participants in this group will receive virtual exercise HIIT training 3 days a week for 12 weeks
  Interventions: Other: HIIT Exercise Training

INTERVENTIONS:
Other: HIIT Exercise Training — The HIIT total session duration will be approximately 30 minutes and will be composed of 10 sets of 60 seconds of high-intensity exercises, >80% of maximum heart rate (MHR), interspersed with a recovery period of 60 seconds of low-intensity exercise at 60% of MHR.

SUMMARY:
The purpose of this study is to compare an onsite to virtual whole-body high intensity interval training (HIIT) program on anthropometric variables, aerobic fitness measures, and vascular markers of cardiac risk in a single study of overweight and obese women.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal adult females over the age of 18 and under the age of 45 with a BMI greater than or equal to 25 and a waist circumference greater than or equal to 35 inches.
* No medical contraindications to participation in an exercise program including major medical illnesses (i.e. cardiovascular disease, stroke, cancer, etc.)
* Ability to provide informed consent
* Willingness and ability to participate in an interval training in-person group fitness exercise program 3x/week for 12 weeks

Exclusion Criteria:

* Adults unable to consent or mini-mental score less than 18.
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Post-menopausal women
* Do not speak English
* Prisoners
* Subjects on medicines (serum glucose, insulin, weight loss medicines, beta-blockers) and having any medical pre-conditions that would interfere with one's capacity to exercise.
* Answer "Yes" to any of the questions on the Pre-Activity Screening Questionnaire (PASQ)

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2021-07-24 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2021-11-08 (Actual)

PRIMARY OUTCOMES:
Pulse Wave Velocity (PWV) | Up to 12 weeks
  vascular marker of cardiac risk will be reported as PWV (m/s) as measured using SphygmoCor
Pulse Wave Analysis Augmentation Index (AIx) | Up to 12 weeks
  vascular marker of cardiac risk will be reported as AIx (%) as measured using SphygmoCor
Pulse Wave Analysis Mean Arterial Pressure (MAP) | Up to 12 weeks
  vascular marker of cardiac risk will be reported as MAP (mmHg) as measured using SphygmoCor
Visceral Adipose Tissue (VAT) content | Up to 12 weeks
  Anthropometric measure will be reported as VAT content as measured by noninvasive direct segmental multi-frequency bioelectrical impedance body composition analyzer
Total Adiposity | Up to 12 weeks
  Anthropometric measure will be reported as Total Adiposity as measured by noninvasive direct segmental multi-frequency bioelectrical impedance body composition analyzer
Aerobic Fitness | Up to 12 weeks
  Aerobic Fitness level as measured by the 20 meter shuttle run

CONTACTS AND LOCATIONS:
Overall Officials: Arlette C Perry, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No